CLINICAL TRIAL: NCT05362903
Title: A Non-interventional Implementation Study to Evaluate Treatment With Inclisiran (Leqvio®) and Other Lipid Lowering Treatments in a Real-world Setting (VICTORION-Implement)
Brief Title: A Non-interventional Implementation Study to Evaluate Treatment With Inclisiran (Leqvio®) and Other Lipid Lowering Treatments in a Real-world Setting
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CKJX839A1DE01
Record Dates: First submitted 2022-04-27; First posted 2022-05-05 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Hypercholesterolemia
Keywords: Hypercholesterolemia; Inclisiran; Atherosclerotic Cardiovascular Disease; ASCVD
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis | interventions — ALN-PCS

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Oral LLT: Patients with documented ASCVD not at individual LDL-C goal and newly initiated on an oral lipid lowering treatment on top of a statin, or alone in patients who are statin-intolerant, or for whom a statin is contraindicated
- Inclisiran: Patients newly initiated on Inclisiran fulfilling the restricted reimbursement criteria or individual access requirements who are not at their individual LDL-C goal as per their CV risk. Two individual sub-cohorts are analysed: 1. Inclisiran in a PCSK9-treatment naive cohort 2. Inclisiran in patients with prior PCSK9 antibody treatment
  Interventions: Other: Inclisiran
- Apheresis plus Inclisiran: Patients who newly initiated Inclisiran on top of lipid apheresis
  Interventions: Other: Inclisiran

INTERVENTIONS:
Other: Inclisiran — Prospective observational cohort study. There is no treatment allocation. Patients administered Inclisiran by prescription will be enrolled.
  Groups: Apheresis plus Inclisiran; Inclisiran

SUMMARY:
This is a multicenter, non-randomized, non-interventional three-cohort study with prospective collection of primary data of treatment with newly initiated oral Lipid lowering treatment on top of a statin (Oral LLT cohort), newly initiated Inclisiran (Inclisiran cohort) and newly initiated Inclisiran on top of lipid apheresis (Apheresis plus Inclisiran cohort) in routine clinical care. All procedures, treatment adaptions and laboratory assessments are part of clinicla routine and conducted independent of this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provide written informed consent to participate in the study
2. Male or female patients ≥ 18 years of age
3. Oral LLT Cohort: Patients with documented ASCVD newly initiated on an oral lipid lowering treatment on top of a statin (e.g. ezetimibe, bempedoic acid, cholestyraimin) or new oral LLT alone in case of statin intolerance or contraindication
4. Inclisiran Cohort: Patients newly initiated on Inclisiran fulfilling the restricted reimbursement criteria or individual access requirements who are not at LDL-C goal as per their CV risk as recommended in the 2019 EAS/ESC guidelines (Mach et al., 2020). At least 60% of the documented patients must be PCSK9-inhibitor naive
5. Apheresis plus Inclisiran Cohort: Patients with Inclisiran on top of regular weekly or bi-weekly lipoprotein apheresis (LDL-c or LP(a)).

Exclusion Criteria:

1. Oral LLT Cohort: Patients who receive a PCSK9-mAB or other PCSK9-targeted therapy
2. Inclisiran 1 Cohort: current or previous PCSK9-targeted treatment
3. Contraindication for Inclisiran according to the SmPC
4. Patients who have received Inclisiran previously
5. Patients with homozygous FH
6. Any underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate) might interfere with interpretation of the clinical study results.
7. Simultaneous or planned participation in an interventional research study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Patients with hypercholesterolemia newly initiated with oral LLT on top of a statin (e.g. ezetimibe, bempedoic acid, cholestyramin), or new oral LLT alone in patients who are statin intolerant (Oral LLT Cohort),
  * Patients newly initiated with Inclisiran according to local reimbursement criteria (out of these, at least 60% naive to monoclonal antibodies targeting PCSK9) (Inclisiran Cohort)
  * Patients treated with Inclisiran on top of lipid apheresis from routine care (Apheresis plus Inclisiran Cohort).
Sampling Method: Non-Probability Sample
Enrollment: 1871 (Actual)
Dates: Start 2022-01-28 (Actual); Primary Completion 2025-11-28 (Actual); Study Completion 2025-11-28 (Actual)

PRIMARY OUTCOMES:
Date of first Atherosclerotic Cardiovascular Disease (ASCVD) diagnosis | Baseline
  Date of first Atherosclerotic Cardiovascular Disease (ASCVD) diagnosis is collected
Number of patients with cardiovascular events | Baseline
  Number of patients with cardiovascular events is collected
Number of participants with concomitant medication in the previous 12 months | Baseline
  Number of participants with concomitant medication in the previous 12 months is collected
Number of apheresis treatments in the previous 12 months | Baseline
  Number of apheresis treatments in the previous 12 months is collected
Lipid lowering therapy used in the previous 12 months | Baseline
  Lipid lowering therapy used in the previous 12 months is collected
Apheresis plus Inclisiran Cohort: Number of lipid apheresis conducted | Baseline
  Number of lipid apheresis conducted on Apheresis plus Inclisiran cohort is collected
Low Density Lipoprotein cholesterol (LDL-C) | Baseline
  Low Density Lipoprotein cholesterol (LDL-C) is collected

SECONDARY OUTCOMES:
Number of In- and outpatient visits | 21 months
  Number of In- and outpatient visits is collected
Number of examinations | 21 months
  Number of examinations is collected
Number and types of lipid lowering treatments | 21 months
  Number and types of lipid lowering treatments are collected
Number of consultations | 21 months
  Number of consultations beside regular visits are collected
Inclisiran Cohort: Percentage of patients progressing to lipoprotein apheresis after initial Inclisiran therapy over time | 21 months
  Percentage of patients progressing to lipoprotein apheresis after initial Inclisiran therapy over time is collected for the Inclisiran Cohort.
Percentage of days covered by at least one LLT | 21 months
  Percentage of days covered (PDC) by at least one lipid lowering treatment (LLT) is collected
Percentage of patients with a PDC ≥ 80% months | 21 months
  Percentage of patients with a Percentage of days covered (PDC) ≥ 80% months is collected
Time to discontinuation of Inclisiran/ any LLT | 21 months
  Time to discontinuation of Inclisiran/ any lipid lowering treatment (LLT) is collected
Percentage of patients who discontinue Inclisiran/ any LLT | 21 months
  Percentage of patients who discontinue Inclisiran/ any lipid lowering treatment (LLT) is collected
Change in LDL-C compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Change in Low denisty lipoprotein cholesterine (LDL-C) compared to baseline is measured
Changes in TC, HDL-C and non-HDL-C compared to Baseline | Baseline, month 3, month 9, month 15, month 21
  Changes in total cholesterol (TC), High Denisty lipoprotein C (HDL-C) and non-HDL-C compared to Baseline is measured
Change in c-reactive protein compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Change in c-reactive protein compared to baseline is measured
Changes in triglycerides and LP(a) compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Changes in triglycerides and Lipoprotein (a) (LP(a)) compared to baseline are measured
Change in hsCRP compared to Baseline | Baseline, month 3, month 9, month 15, month 21
  Change in high-sensitivity C-reactive protein (hs-CRP) compared to Baseline is measured
Change in Creatinin compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Change in Creatinin compared to baseline is measured
Change in HbA1c compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Change in Glycated hemoglobin (HbA1c) compared to baseline is measured
Change in eGFR compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Change in Estimated Glomerular Filtration Rate (eGFR) compared to baseline is measured
Proportion of patients achieving prespecified LDL-C targets | Baseline, month 3, month 9, month 15, month 21
  Proportion of patients achieving prespecified LDL-C targets based on 2019 ESC/EAS guideline for the management of dyslipidemia is collected
Percentage of patients achieving ≥50% LDL-C reduction over time | Baseline, month 3, month 9, month 15, month 21
  Percentage of patients achieving ≥50% LDL-C reduction over time is collected
Changes in SMART-Risk Scores over time compared to baseline | Baseline, month 3, month 9, month 15, month 21
  The SMART Risk Score is a tool to estimate 10-year risk for recurrent vascular events in patients with manifest cardiovascular disease. SMART Risk Score ranges from 0 - 100 %, where higher values indicate higher cv risk.
Proportion of patients with treatment modifications | 21 months
  Proportion of patients with the following treatment modifications, is collected:
  * dose changes
  * switching of lipid lowering treatment
  * initiation of lipid apheresis for LDL-C
Changes from baseline in WHO Quality of Life BREF (WHOQOL-BRED)questionnaire over time | Baseline, month 3, month 9, month 15, month 21
  Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed linearly to a 0-100-scale. Higher numbers indicate better QoL.
Changes from baseline in TSQM-9 over time | Baseline, month 3, month 9, month 15, month 21
  Treatment Satisfaction Questionnaire for Medication-9 items (TSQM-9) domain scores range from 0 -100, with higher scores representing higher satisfaction on that domain.
Evaluate nutritional factors via questionnaire | Baseline, month 3, month 9, month 15, month 21
  Questionnaire from the German "Nationale Verzehrstudie II -Was esse ich" is used. No score is used for the interpretation. Questions about nutrition and activities are interpreted separately and compared over time.
Percentage of Adverse Events and Serious Adverse Events | 21 months
  Percentage of Adverse Events (AEs) and Serious Adverse Events (SAEs) is collected
Percentage of Adverse Events and Serious Adverse Events leading to discontinuation of therapy | 21 months
  Percentage of Adverse Events and Serious Adverse Events leading to discontinuation of therapy is collected
Apheresis plus Inclisiran Cohort: Changes in the rate of lipid apheresis | 12 months pre-Baseline, Baseline, month 3, month 9, month 15, month 21
  Changes in the rate of lipid apheresis over time after Inclisiran initiation compared to the period 12 months pre-Baseline is collected.
Apheresis plus Inclisiran Cohort: Changes in CRP compared to baseline | Baseline, month 3, month 9, month 15, month 21
  Changes in high-sensitive C-reactive protein (hsCRP) are measured in labs. Values are interpresetd as;
  - less or 1.0 mg/l is normal 1.01 - 3.00 slightly high more than 3.0 mg/l is significantly elevated
Apheresis plus Inclisiran Cohort: Changes in PTH | Baseline, month 3, month 9, month 15, month 21
  Apheresis plus Inclisiran Cohort: Changes in Parathyroid hormone (PTH)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (103):
- Germany (103):
  - Novartis Investigative Site, Freudenstadt, Baden-Wurttemberg
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Kirchheim unter Teck, Baden-Wurttemberg
  - Novartis Investigative Site, Konstanz, Baden-Wurttemberg
  - Novartis Investigative Site, Coburg, Bavaria
  - Novartis Investigative Site, Dachau, Bavaria
  - Novartis Investigative Site, Deggendorf, Bavaria
  - Novartis Investigative Site, Füssen, Bavaria
  - Novartis Investigative Site, Grünwald, Bavaria
  - Novartis Investigative Site, Landshut, Bavaria
  - Novartis Investigative Site, Marktoberdorf, Bavaria
  - Novartis Investigative Site, Muehldorf Am Inn, Bavaria
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Burg, Brandenburg
  - Novartis Investigative Site, Potsdam, Brandenburg
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Rotenburg (Wümme), Lower Saxony
  - Novartis Investigative Site, Winsen, Lower Saxony
  - Novartis Investigative Site, Stralsund, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Detmold, North Rhine-Westphalia
  - Novartis Investigative Site, Mülheim, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Ingelheim, Rhineland-Palatinate
  - Novartis Investigative Site, Kaiserslautern, Rhineland-Palatinate
  - Novartis Investigative Site, Chemnitz, Saxony
  - Novartis Investigative Site, Eberswalde, Saxony
  - Novartis Investigative Site, Görlitz, Saxony
  - Novartis Investigative Site, Hohenstein-Ernstthal, Saxony
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Pirna, Saxony
  - Novartis Investigative Site, Halle, Saxony-Anhalt
  - Novartis Investigative Site, Quedlinburg, Saxony-Anhalt
  - Novartis Investigative Site, Greiz, Thuringia
  - Novartis Investigative Site, Jena, Thuringia
  - Novartis Investigative Site, Siegen, Westfalia
  - Novartis Investigative Site, Lutherstadt Witten, Wittenberg
  - Novartis Investigative Site, Altenburg
  - Novartis Investigative Site, Aue
  - Novartis Investigative Site, Bad Homburg
  - Novartis Investigative Site, Bad Nauheim
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Biedenkopf
  - Novartis Investigative Site, Borsdorf
  - Novartis Investigative Site, Brilon
  - Novartis Investigative Site, Brüel
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Cloppenburg
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Cuxhaven
  - Novartis Investigative Site, Dachau
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Dessau
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Ehingen
  - Novartis Investigative Site, Ehringshausen
  - Novartis Investigative Site, Eisfeld
  - Novartis Investigative Site, Frechen
  - Novartis Investigative Site, Fürth
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Günzburg
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Heide
  - Novartis Investigative Site, Hennigsdorf
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, Markkleeberg
  - Novartis Investigative Site, Moers
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Naumburg
  - Novartis Investigative Site, Neumarkt
  - Novartis Investigative Site, Neuruppin
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Offenbach
  - Novartis Investigative Site, Olpe
  - Novartis Investigative Site, Oranienburg
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Osnabrück
  - Novartis Investigative Site, Papenburg
  - Novartis Investigative Site, Pirmasens
  - Novartis Investigative Site, Rendsburg
  - Novartis Investigative Site, Riesa
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Salzatal
  - Novartis Investigative Site, Schwandorf in Bayern
  - Novartis Investigative Site, Schwedt
  - Novartis Investigative Site, Speyer
  - Novartis Investigative Site, Stadtlohn
  - Novartis Investigative Site, Trier
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Wermsdorf
  - Novartis Investigative Site, Wesel
  - Novartis Investigative Site, Winterberg
  - Novartis Investigative Site, Wismar
  - Novartis Investigative Site, Wuppertal
  - Novartis Investigative Site, Würzburg
  - Novartis Investigative Site, Zwiesel

IPD SHARING:
Plan to Share IPD: No